CLINICAL TRIAL: NCT02664311
Title: A Randomized Comparison of the Use of JET and Conventional Ventilation in Pulmonary Vein Isolation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: under enrollment
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Alfred Buxton, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2012P000419
Record Dates: First submitted 2014-09-24; First posted 2016-01-27 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
Keywords: Pulmonary Vein Isolation; Jet Ventilation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — High-Frequency Jet Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Ventilation (Placebo Comparator): Patients receiving conventional ventilation for the duration of this study
  Interventions: Device: Conventional ventilation
- Jet Ventilation (Active Comparator): Patients receiving Jet ventilation while under general anesthesia and during mapping and ablation in the left atrium
  Interventions: Device: Jet Ventilation

INTERVENTIONS:
Device: Jet Ventilation — Patients are randomized to receive either jet or conventional ventilation during this study
  Arms: Jet Ventilation
Device: Conventional ventilation — Conventional ventilator - control arm
  Arms: Conventional Ventilation

SUMMARY:
This is a randomized prospective study comparing outcomes of pulmonary vein isolation using conventional and jet ventilation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia in the United States today. Its incidence increases with age, and the prevalence approaches 10% in patients over 80 years old. Atrial fibrillation increases the risk of strokes, and in some patients is associated with worsened congestive heart failure and quality of life.

Catheter based radiofrequency ablation for atrial fibrillation is an evolving and promising technology, and provides increased freedom from AF and improved quality of life compared with pharmacologic therapy. The technique involves placing catheters through the femoral veins into the heart, including the left atrium. Access to the left atrium is performed by transseptal puncture. Ablation of atrial fibrillation is performed by delivery of radiofrequency energy around the pulmonary veins in order to electrically dissociate them from the atria. This is thought to eliminate common triggers for atrial fibrillation, and therefore reduces the recurrence of AF in some patients.

The ablation procedure is done under general anesthesia and takes 4-8 hours. The first part of the procedure involves creating a computer generated three dimensional model of the left atrium. Once this model is created any patient movement will disrupt its accuracy and interfere with the physician's ability to accurately locate the catheter within the atrium.

The success of AF ablation is dependent upon the creation of an accurate three dimensional model, as well as physicians ability to perform durable lesions and achieve effective isolation of the pulmonary veins. Among the barriers to technical success are the patient's respiratory movement, which impairs catheter stability and the ability to maintain a stable catheter position against the atrium of the heart during ablation. Thus, minimizing respiratory movement during the procedure is critical to procedural outcome.

High frequency jet ventilation (HFJV) is a newer mode of ventilation that relies on very small tidal volumes delivered at high frequency (approximately 80-120 breaths/minute). Initially developed in the critical care setting, HFJV produces less respiratory motion due the small tidal volumes delivered. HFJV has been used successfully in procedures requiring increased stability of the field of interest, such as lithotripsy and percutaneous hepatic and renal radiofrequency ablation as well as stereotactic high single-dose irradiation of stage I non-small cell lung cancer and lung metastases. The initial report of the use of HFJV in radiofrequency catheter ablation (RFCA) of atrial fibrillation was by Goode et al in 2006. In that retrospective analysis, the use of HFJV was associated with a decrease in the number of ablation lesions, due to decreased number of attempts aborted by catheter dislodgement, as well as decreased variation in the size of the left atrium (LA) due to changes in pulmonary pressures associated with conventional ventilation. The incidence of complications was not significantly different between the HFJV and conventionally ventilated patients. More recently, Elkassabany et al. retrospectively reviewed their institutional experience with Jet ventilation, and found that the procedure could be performed safely.

HFJV is increasingly used and may improve procedure efficacy and safety, and may be cost effective. Data however are limited to small series and retrospective reviews. In order to better compare the efficacy and safety of HFJV to conventional ventilation, the investigators propose to conduct a prospective randomized study comparing the use of HJFV and conventional ventilation in patients undergoing pulmonary vein isolation (PVI) at our institution. Our hypothesis is that HFJV, by allowing greater catheter stability and more accurate mapping of the left atrium will allow more effective radiofrequency lesion creation, leading to a quicker procedure, requiring fewer lesions and less ablation and fluoroscopy time with more effective isolation of the pulmonary veins with better short and long term control of AF.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal or persistent AF, first time PVI or left atrial procedure

Exclusion Criteria:

* repeat procedure
* any contraindications to receiving JET ventilation in the judgement of the treating anesthesiologist

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zimetbaum, MD, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication in scientific journal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2013-January 2014 at Beth Israel Deaconess Medical Center
Period: Overall Study
Arm/Group | Conventional Ventilation | Jet Ventilation
Started | 6 | 3
Completed (Insufficient faculty interest to recruit patients) | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Ventilation | Jet Ventilation | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (17) | 60 (9) | 59 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9
Atrial fibrillation [Count of Participants; unit: Participants]
  Atrial fibrillation - paroxysmal | 4 | 1 | 5
  Atrial fibrillation - persistent | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Isolation Time
Description: Comparison of Time (in Minutes) From Obtaining Access to Left Atrium Via Transseptal Catheterization to Demonstrated Isolation of All Pulmonary Veins - hypothesis is that with Jet ventilation there will be a shorter time to pulmonary vein isolation in comparison to conventional ventilation
Time Frame: Immediate post procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Conventional Ventilation | Jet Ventilation
Number analyzed (Participants) | 6 | 3
minutes | 127 (45) | 117 (55)

2. Secondary Outcome: Freedom From AF
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Ventilation | Jet Ventilation
Number analyzed (Participants) | 6 | 3
Participants | 6 | 3

3. Secondary Outcome: Fluoroscopy Time
Description: Fluoro time as recorded by RNs from Xray machine
Time Frame: Immediate post-procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Conventional Ventilation | Jet Ventilation
Number analyzed (Participants) | 6 | 3
minutes | 54 (11.9) | 48 (18.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Conventional Ventilation | Jet Ventilation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No